CLINICAL TRIAL: NCT00410501
Title: An Open Label, Single Dose, Two Period, Single Sequence Crossover Study to Assess the Pharmacokinetic Interaction of QAB149 (300 Mcg Via Inhalation) With Ketoconazole (200 mg Tablet b.i.d.) in Healthy Adult Subjects
Brief Title: Evaluation of Pharmacokinetic Interaction of Indacaterol With Ketoconazole in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149A2311
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics, interaction, QAB149, indacaterol, ketoconazole, healthy subjects
MeSH Terms: interventions — indacaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Indacaterol (QAB149)

SUMMARY:
This study will evaluate the interaction potential between indacaterol and ketoconazole (a potent CYP3A inhibitor) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects of Indian origin age 18 to 45 years of age (inclusive)
* In good health as confirmed by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis on the screening and baseline evaluation
* Female subjects must be either surgically sterilized at least 6 months prior to study participation or post-menopausal (no regular menstrual bleeding for at least 2 years), or using a double-barrier local contraception if of childbearing potential
* Body mass index (BMI) within the range of 18.5 to 27 kg/m2 and weigh at least 45 kg for females and 50 kg for males

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months).
* Using or planning to use medications affecting GI (gastrointestinal) motility and/or perception (prokinetics, antidiarrheals, antispasmodics, anticholinergics, antacids containing magnesium or aluminum salts, erythromycin, octreotide, ondansetron or other 5-HT3 antagonists).
* Use of any prescription drugs within 4 weeks prior to dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within two (2) weeks prior to dosing. Paracetamol (up to 4 g daily) is acceptable
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* A past medical history of clinically significant ECG abnormalities. Significant history of psychiatric disorder.
* History of clinically significantfainting, low blood pressure when standing, irregular heart beats or acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or untreated) drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis, nasal polyp or NSAID (non-steroidal anti-inflammatory drug) induced urticaria)
* A known hypersensitivity or severe adverse event to indacaterol/ketoconazole or drugs similar to the study drugs.
* History of bowel obstruction, symptomatic gall bladder disease, suspected Sphincter of Oddi dysfunction, or abdominal adhesions.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* Any planned surgery or procedure within 3 months of screening.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C or VDRL (Venereal Disease Research Laboratory) test result.
* History of drug or alcohol abuse within the 6 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations. Consumption of alcohol within 48 hours of receiving medication.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-12

PRIMARY OUTCOMES:
Pharmacokinetics of a single 300 µg dose of indacaterol (QAB149) alone administered via inhalation and in the presence of ketoconazole (at steady state) in healthy adult subjects

SECONDARY OUTCOMES:
Safety of a single 300 µg dose of indacaterol (QAB149) given via inhalation in the presence of ketoconazole at steady state in healthy adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Investigator site
Locations (1):
- Novartis, Mumbai, India